CLINICAL TRIAL: NCT05082974
Title: A Randomized, Controlled, Double-Masked, Two-Arm Investigator-Initiated Study to Assess the Efficacy of OC-01 (Varenicline) Nasal Spray on Signs and Symptoms of Dry Eye Disease in Subjects Following Laser-assisted in Situ Keratomileusis (LASIK)
Brief Title: Investigator Initiated Study to Assess the Efficacy of OC-01 (Varenicline) Nasal Spray on Signs and Symptoms of Dry Eye Disease Following Laser-assisted in Situ Keratomileusis (LASIK)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vance Thompson Vision ND (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: The RANK Study
Record Dates: First submitted 2021-10-05; First posted 2021-10-19 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Dry Eye Disease
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Varenicline; Nasal Sprays

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- OC-01 (varenicline 0.6mg/ml) nasal spray (Experimental)
  Interventions: Drug: OC-01 (varenicline 0.6mg/ml) nasal spray
- Placebo (vehicle) nasal spray (Placebo Comparator)
  Interventions: Drug: Placebo (vehicle) nasal spray

INTERVENTIONS:
Drug: OC-01 (varenicline 0.6mg/ml) nasal spray — OC-01 (varenicline 0.6mg/ml) nasal spray which contains varenicline is being developed by Oyster Point Pharma for the treatment of signs and symptoms of Drye Eye Disease. OC-01 (varenicline) nasal spray activates the trigeminal parasympathetic pathway and stimulates natural tear production to bathe the corneal nerve endings in a protective layer of tear film. In addition, OC-01 (varenicline) acts as a cholinergic agonist and may provide analgesia by activating the trigeminal parasympathetic pathway.
  Arms: OC-01 (varenicline 0.6mg/ml) nasal spray
Drug: Placebo (vehicle) nasal spray — Placebo (vehicle) nasal spray [control]
  Arms: Placebo (vehicle) nasal spray

SUMMARY:
Evaluate the safety and effectiveness of OC-01 (varenicline) nasal spray for amelioration of signs and symptoms of dry eye disease in subjects following laser-assisted in situ keratomileusis (LASIK).

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to sign the informed consent form (ICF)
* Be at least 18 years of age at the screening visit
* Be undergoing LASIK treatment in one or both eyes
* Be myopic between -1.00D to -7.00D MRSE (manifest refraction spherical equivalent) in study eye (right eye) with ≤2D between eyes or subjects undergoing monovision treatment with study eye (distance eye) meeting the diopter requirement of myopia
* Be literate and able to complete questionnaires independently
* Be able and willing to use the study drug and participate in all study assessments and visits
* Have sufficient hand strength, in the opinion of the Investigator, to be able to independently administer the study drug
* Have provided verbal and written informed consent
* If a female is of childbearing potential, they must: use an acceptable means of birth control (acceptable methods of contraception include: hormonal - oral, implantable, injectable, or transdermal contraceptives, mechanical - spermicide in conjunction with a barrier such as a diaphragm or condom, IUD, or surgical sterilization of partner), and have a negative urine pregnancy test on baseline

Exclusion Criteria:

Subjects must not:

* Have a break in the integrity of the corneal epithelium such as a persistent corneal epithelial defect, or corneal ulcer.
* Have presence of corneal pathology that may interfere with LASIK outcomes
* Active infectious, ocular or systemic disease
* Have a history of ocular inflammation or macular edema
* Have had clinically significant active infectious keratitis in the past 3 months
* Have history of prior refractive surgery
* Have placement of temporary punctal plugs in the past 1 month or current presence of permanent punctal plugs at time of screening
* Have chronic or recurrent epistaxis, coagulation disorders or other conditions that, in the opinion of the Investigator, may lead to clinically significant risk of increased bleeding
* Have had nasal or sinus surgery (including history of application of nasal cautery) or significant trauma to these areas
* Have a vascularized polyp, severely deviated septum, chronic recurrent nosebleeds, or severe nasal obstruction as confirmed by intranasal examination performed at Visit 1.
* Be currently treated with nasal continuous positive airway pressure
* Have had blepharoplasty in either eye
* Have had a corneal transplant in either eye
* Have a history of seizures or other factors that lower the subject's seizure threshold.
* Have a systemic condition or disease not stabilized or judged by the Investigator to be incompatible with participation in the study or with the lengthier assessments required by the study (e.g., current systemic infection, uncontrolled autoimmune disease, uncontrolled immunodeficiency disease, history of myocardial infarction or heart disease, etc.)
* Have a known hypersensitivity to any of the procedural agents or study drug components
* Have current concomitant use of a nicotinic acetylcholine receptor agonist [Nicoderm®, Nicorette®, Nicotrol NS® (nicotine), Tabex®, Desmoxan® (cytisine), and Chantix® (varenicline)] within the previous 30 days of Visit 1 and during the treatment period.
* Have current concomitant use of snuff, chewing tobacco, e-cigarettes or cigarettes/cigars during the study or within the previous 30 days.
* Subject must refrain from smoking during the course of the study.
* Have active or uncontrolled, severe at the discretion of the investigator:

  * Systemic allergy
  * Chronic seasonal allergies at risk of being active during the study treatment period
  * Rhinitis or sinusitis requiring treatment such as antihistamines, decongestants, oral or aerosol steroids at the Screening Visit or be expected to require treatment during the treatment period of the study
* Untreated nasal infection at Visit 1
* Have any condition or history that, in the opinion of the investigator, may interfere with study compliance, outcome measures, safety parameters, and/or the general medical condition of the subject
* Be currently enrolled in an investigational drug or device study or have used an investigational drug or device within 30 days prior to Visit 1 and during the treatment period.
* Be a female who is pregnant, nursing, or planning a pregnancy at Visit 1. Be a woman of childbearing potential who is not using an acceptable means of birth control; acceptable methods of contraception include: hormonal - oral, implantable, injectable, or transdermal contraceptives; mechanical - spermicide in conjunction with a barrier such as a diaphragm or condom; IUD; or surgical sterilization of partner or hysterectomy. A woman that has not had a menses in 12 months or longer is not considered of childbearing potential.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-10-20 (Actual); Primary Completion 2022-08-03 (Actual); Study Completion 2022-08-03 (Actual)

PRIMARY OUTCOMES:
Change in NEI-VFQ-25 (National Eye Institute Visual Function Questionnaire) score | Baseline to Day 84 (3 months)
  25 questions to determine overall score of dry eye disease symptoms completed by subject. Scored from 0-100, with 100 being the highest score and best outcome.
Mean change in corneal fluorescein staining based on the NEI (National Eye Institute) scale for Corneal Fluorescein Staining determined at slit lamp | Baseline to Surgical Day and from Surgical Day to Day 84 (3-month)
  Evaluated at slit lamp by a masked physician

SECONDARY OUTCOMES:
Change in NEI-VFQ-25 (National Eye Institute Visual Function Questionnaire) score | Baseline to Day 184 (6 months)
  25 questions to determine overall score of dry eye disease symptoms completed by subject. Scored from 0-100, with 100 being the highest score and best outcome.
Mean change in eye dryness score (EDS) | Baseline to Day 184 (6 months)
  Eye dryness score (EDS) measured by the Visual Analogue Scale (VAS). Scored from 0-100, with 100 being the worst pain imaginable, and zero no pain.
Mean change in residual refractive error | Day 28 (1-month) postoperative LASIK over time to Day 84 (3-month) postoperative LASIK
  Evaluated by manifest refraction
Change in tear collection lab values | Day 28 (1-month) postoperative LASIK over time to Day 84 (3-month)
  As determined by Schirmer's strips
Mean change tear break-up time | baseline to Day 0 (Surgical Day), Day 28 (1-month) postoperative LASIK and Day 84 (3-month) postoperative LASIK
  As determined by tear break-up testing
Proportion of subjects treated with rescue dry treatment and/or punctal plugs | Day 84 (3-months) postoperative and Day 168 (6-months) postoperative LASIK
  Determined at follow up appointment by Doctor
Incidence and severity of adverse events | Screening to Day 168 (6-month postoperative LASIK)
  As reported by study coordinators and evaluated by PI

CONTACTS AND LOCATIONS:
Locations (1):
- Vance Thompson Vision ND, West Fargo, North Dakota, United States